CLINICAL TRIAL: NCT04616235
Title: Acute Exercise and NK Cell Regulation in Tissue and Circulation After IL-6R Blockade - a Randomized Controlled Trial
Brief Title: Acute Exercise and NK Cell Regulation in Tissue and Circulation After IL-6R Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Andreas Kraag Kraag Ziegler, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: jr. nr. H-20028611
Record Dates: First submitted 2020-10-20; First posted 2020-11-04 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Interleukin-6 Inhibition; Physical Stress; Appetitive Behavior
Keywords: Natural Killer cells; Aerobic exercise; IL-6R blockade; Human; Appetite
MeSH Terms: conditions — Appetitive Behavior | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The IL-6R receptor blockade infusion will have bag concealment so that neither the scientific staff or the subject will know if Tocilizumab or saline (placebo) is given and we do not expect the subjects to "feel" the infusion or the results of the infusion.
  All scientific staff will be blinded to group allocation using encryption. Only once all data have been obtained (histology, blood analysis, gene-expression, Western Blot, Flow cytometry, single cell RNA sequencing) concealment will be broken so that statistical analysis can be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CON (Placebo Comparator): This group will do intense aerobic exercise without concomitant IL-6R blockade
  Interventions: Other: Saline 0.9% 100 ml NaCl 0.9% will be infused over 1 hour
- BLOCK (Active Comparator): This group will do intense aerobic exercise with concomitant IL-6R blockade
  Interventions: Drug: Tocilizumab Injectable Product

INTERVENTIONS:
Drug: Tocilizumab Injectable Product — The intervention group will undergo intense aerobic exercise with prior IL-6R infusion for 1h prior to the exercise bout.
  Arms: BLOCK
Other: Saline 0.9% 100 ml NaCl 0.9% will be infused over 1 hour — The control group will undergo intense aerobic exercise with saline infusion for 1h prior to the exercise bout
  Arms: CON

SUMMARY:
The study is a randomized controlled trial studying the acute effect of intense aerobic exercise upon NK (Natural Killer) cell activation and appetite-regulation in human participants with or without concommitant IL-6R receptor blockade (Tocilizumab)

DETAILED DESCRIPTION:
Objectives:

Primary Objective:

* To explore the association between acute exercise, IL-6 blockade and NK regulation in circulation.
* To explore whether exercise activated NK-cells have a unique phenotype using single cell RNA sequencing.

Secondary Objectives:

* To explore the effect of acute aerobic exercise on NK cell number and activity in circulation, muscle and adipose tissue, in healthy young males, in order to indirectly explore exercise as an anti-cancer remedy.
* To assess the kinetics of the NK-cell response and, if possible, chronologically investigate the appearance and whereabouts of the activated NK-cells.

Explorative Objectives

* To establish a reproducible protocol for tracking various immune-cells and their involvement in the acute exercise response in humans
* To investigate novel signal molecules released from muscle during exercise with immunological importance.
* To investigate the possible role of exercise induced IL-6 on subjective feelings of hunger and satiety post exercise and food intake. • To explore the effect of IL-6 receptor blockade on the exercise proteome and metabolome, using mass spectrometry

Methods:

30 healthy recreationally active young males will be included in this acute exercise study in which NK-cell kinetic and regulation will be studied in response to acute aerobic exercise and IL-6R blockade or placebo.

The study consists of 2 visits. At inclusion (visit 1) all subjects will undergo assessment encompassing: baseline medical screening (auscultation, blood pressure, ECG), determination of body composition (DXA), cardiovascular fitness (VO2max) and standard fasting blood-biochemistry which will be analyzed immediately. Visit 2 will consist of a muscle and fat biopsy from the dominant leg and abdominal subcutaneous-fat depot respectively (both under resting conditions), which will then act as reference tissue for the further tissue analysis. Then, a 18G antecubital peripheral venous access will be secured prior to commencing with IL-6R infusion. 2 hours after the infusion procedure the subjects will undergo an acute exercise protocol. Subjects will then be challenged by a high intensity acute aerobic exercise bout, utilizing a bicycle ergometer. Blood samples will be drawn prior to the infusion and exercise, during exercise, as well as immediately, ½, 1, 1½ and 2h post exercise and up 4h post exercise in the appetite regulation substudy. Blood samples will immediately be analyzed for leucocyte count and differentiation as well as plasma biochemistry. In addition, blood samples will be utilized for NK cell isolation with subsequent single cell RNA sequencing, immune cell distribution and killing capacity towards cancer cells. Furthermore, plasma samples will be collected and frozen for later determination of cortisol, prolactin and circulating cytokines, including but not limited to IL-6 and G-CSF. Lastly, in the appetite substudy, insulin, GLP-1 and free fatty acids will be measured.

Tissue samples will be obtained 2h post exercise for optimizing gene-expression analysis. Both muscle and adipose tissue samples will be analyzed for inflammatory and anti-inflammatory markers, NK cell content and phenotyping of these NK cells using markers obtained from single cell sequencing, conducted on the blood-borne NK-cells. Furthermore, immune cell infiltration will be assessed using histology. All tissue samples will be obtained using a Bergström needle under sterile conditions during local anesthesia in order to minimize any sample-related discomfort or infection.

After the tissue sample, an ad libitum meal will be served, the subjects can eat as much can, but are instructed not to overconsume as any leftover food can be taken home. Paracetamol (1.5g) will be given to asses gastric emptying.

All participants will undergo the 2 study visits at the same approximate time of the day (9.00 a.m.) After completion of the study, any left-over material will be transferred to the CFAS biobank.

Subjects: Included subjects will be 30 recreationally active, moderately trained, healthy young males aged 18-40 years. Exclusion criteria are: cardiovascular, rheumatologic and metabolic disease, elite sports or high aerobic training status. Chronic use of nonsteroidal anti-inflammatory drug (NSAID) or other immunosuppressants.

Intervention: Subjects will be randomized to acute exercise, with (n=15) or without (n=15) prior IL-6R blockade. The exercise intervention will consist of a highly taxing ≈45 minutes interval based, aerobic exercise bout, conducted on a stationary bicycle ergometer. After an initial 5-minute warmup at 50-60% of HRmax, subjects will undergo seven, verbally encouraged, 3-minute intervals at above 90% HRmax, interspersed by 3 minutes of low intensity pedaling. Blood samples will be drawn before, during as well as immediately, ½, 1, 1½ and 2h post exercise together with tissue sampling at the 2h time-point.

To assess appetite regulation, further blood samples will be drawn from 2h-4h post exercise.

Statistical considerations: Based on data from our pilot study, we anticipate a ≈ 45 % lower maximal NK cell mobilization in the IL6R inhibition group compared to CON and a 29 % difference in NK cell nadir with the lowest values obtained in the IL6R inhibition group. Assuming a 5%-significance level in two-sided tests, we need to include 9 patients in each group to achieve 90% power for detecting a relative difference of 45 % in the intervention-group. To account for potential dropouts/excluded, due to the somewhat invasive setup, we will include a total of 30 patients (15 per group).

Recruitment: Subjects will be recruited through forsøgsperson.dk or similar sites alongside advertising at relevant sites.

Subjects will contact us at CFAS and will be given the choice whether to receive study information pr. telephone (thereby denying the option of a bystander) or a face to face meeting at CFAS. All this information will be given by the primary investigator. If the subject is interested in hearing more of the study, relevant documents will be emailed. If the subject is interested in joining the study after having received written or oral information, he will have 24h to consider study participation. When the subject has been informed either by telephone or face to face and accepts study participation, he will be invited to visit 1 where written and informed consent will be obtained (or signed and brought from home by the participant).

Risks and adverse reactions: Subjects may experience minor discomfort with regard to blood and tissue samples. The blood volume drawn is negligible and will not be associated with any health risk. All sampling of tissues will be performed under sterile conditions during local anesthesia and will thus be associated with little pain or discomfort and very little risk of infection. During exercise testing, participants may experience shortness of breath.

IL-6R inhibition is generally well tolerated with only few side-effects. The dose of paracetamol is low and is not associated with any risk.

Contact information of the involved medical doctor will be given to participants at study inclusion, so that any adverse event can be reported and solved.

Dissemination of study results: Both positive, negative and inconclusive results will be published in relevant international scientific journals.

Ethical consideration: The project is expected to cause limited risks, side effects and discomfort. All procedures will be performed by experienced physicians and physiologists with relevant safety. Tocilizumab is generally well tolerated and the dose of paracetamol is low. Included subjects may at any time, and without justification, retract their consent of study participation. We believe that the project is important and will contribute with critical new information on the IL-6 modifiable NK-cell response to acute exercise both in circulation and in adipose and muscle tissue (as there is currently very limited knowledge on the latter).

The study is considered a toolbox-study by Lægemiddelstyrelsen, and hence not at pharmaceutical study

ELIGIBILITY:
Inclusion Criteria:

* recreationally active
* moderately trained
* healthy young males aged 18-40 years
* BMI from 18-30 kg·m2

Exclusion Criteria:

* Cardiovascular disease
* Rheumatologic disease
* Metabolic disease,
* Elite sports or high aerobically training status (VO2max>60ml O2/min/kg),
* Frequent/chronic use of medications affecting physical performance or inflammation (NSAIDS, DMARDS)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants will have to be biological males since hormonal fluctuations in women might have unknown effects on immune cell regulation during acute intense exercise
Enrollment: 30 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Kinetics and regulation of NK (Natural Killer) cells during and following acute exercise | Up to 1 day
  Change in NK cell and NK cell subset count in circulation before and after acute aerobic exercise with or without IL-6R blockade.
NK cell phenotype in response to acute exercise with or without IL-6R blockade | Up to 1 day
  Change in NK-cell phenotype using single cell RNA sequencing. Here, within-group changes of baseline vs. post exercise timepoints as well as between group differences between IL-6 blockade and placebo will be investigated.
  The focus will be on markers of cytotoxicity, cell adhesion and adrenergic signaling.

SECONDARY OUTCOMES:
Change in NK cell count in adipose tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD56, CD57 and other NK-cell markers, the principal investigator will identify and count the number of NK cells in adipose tissue
Change in NK cell phenotype in adipose tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD56, CD57 and other NK-cell markers, the principal investigator will identify the phenotype of NK cells in adipose tissue
Change in NK cell count in muscle tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD56, CD57 and other NK-cell markers, the principal investigator will identify and count the number of NK cells in muscle tissue
Change in NK cell phenotype in muscle tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD56, CD57 and other NK-cell markers, the principal investigator will identify the phenotype of NK cells in muscle tissue
Change in macrophage count in muscle tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD68, CD163, CD206, TNF-alpha and other macrophage markers, the principal investigator will identify and count the number of macrophages in muscle tissue
Change in macrophage phenotype in muscle tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD68, CD163, CD206, TNF-alpha and other macrophage markers, the principal investigator will phenotype (M1/M2) macrophages in muscle tissue
Change in macrophage count in adipose tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD68, CD163, CD206, TNF-alpha and other macrophage markers, the principal investigator will identify and count the number of macrophages in adipose tissue
Change in macrophage phenotype in adipose tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD68, CD163, CD206, TNF-alpha and other macrophage markers, the principal investigator will phenotype (M1/M2) macrophages in adipose tissue
Change in T-cell count in adipose tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD3, CD8, and other T-cell markers, the principal investigator will count the number of T-cells in adipose tissue
Change in T-cell phenotype in adipose tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD3, CD8, and other T-cell markers, the principal investigator will phenotype the T-cells in adipose (CD3+/CD8+) tissue
Change in T-cell count in muscle tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD3, CD8, and other T-cell markers, the principal investigator will count the number of T-cells in muscle tissue
Change in T-cell phenotype in muscle tissue | 3 hours after intervention
  Using a combination of histology, western blot and gene-expression analysis for CD3, CD8, and other T-cell markers, the principal investigator will phenotype (CD3+/CD8+) the T-cells in muscle tissue
Change in monocyte count in circulation | Up to 1 day
  Using flow cytometry we will identify and count monocytes in circulation
Change in T-cell count in circulation | Up to 1 day
  Using flow cytometry the investigators will count T-cells in circulation
Change in B-cell count in circulation | Up to 1 day
  Using flow cytometry the investigators will count B-cells in circulation
Change in IL-6 receptor expression on NK-cells in circulation | Up to 1 day
  The change in IL-6 receptor surface expression on circulating NK-cells using flow cytometry
Change in circulating IL-6 | Up to 1 day
  Plasma IL-6 conc. using ELISA assay
Change in circulating IL-2 | Up to 1 day
  Plasma IL-2 conc. using ELISA assay
Change in circulating IL-1 | Up to 1 day
  Plasma IL-1 conc. using ELISA assay
Change in circulating IL-10 | Up to 1 day
  Plasma IL-10 conc. using ELISA assay
Change in circulating TNF-alpha | Up to 1 day
  Plasma TNF-alpha conc.using ELISA assay
Change in circulating G-CSF | Up to 1 day
  Plasma TNF-alpha conc. using ELISA assay
Change in circulating epinephrine | Up to 1 day
  Blood epinephrine conc. using ELISA assay
Change in circulating norepinephrine | Up to 1 day
  Blood norepinephrine conc. using ELISA assay
Change in circulating total leucocytes | Up to 1 day
  Blood leucocyte count using sysmex XN
Change in circulating neutrophils | Up to 1 day
  Blood neutrophil count.using sysmex XN
Change in circulating reticulocytes | Up to 1 day
  Blood reticulocytes count.using sysmex XN
Change in circulating eosinophils | Up to 1 day
  Blood eosinophil count.using sysmex XN
Change in circulating basofile leucocytes | Up to 1 day
  Blood basofile leucocytes count.using sysmex XN
Change in circulating total lymphocytes | Up to 1 day
  Blood lymphocyte count.using sysmex XN
Change in circulating Prolactin | Up to 1 day
  Plasma Prolactin conc. using sysmex XN
Change in cortisol | Up to 1 day
  Plasma cortisol conc. using sysmex XN
Change in metamyelocytes | Up to 1 day
  Blood metamyelocyte count using sysmex XN
Change in ACTH | Up to 1 day
  Plasma ACTH conc. using sysmex XN
Change in circulating lactate | Up to 1 day
  Blood lactate using ABL
Change in CRP | Up to 1 day
  Plasma CRP conc. using sysmex XN
Change in hsCRP | Up to 1 day
  Plasma CRP conc. using ELISA
Novel myokines during acute exercise | Immediately after acute bout of exercise
  As an explorative outcome the investigators will investigate possible novel signal molecules released during exercise with immunological importance, either in circulation or in tissue (i.e. GDNF [Glial cell Derived Neurotrophic Factor])
VO2max | Baseline
  VO2max using bicycle ergometer and Oxicon Online system
Lean Body mass | Baseline
  Lean body mass using dual-energy x-ray absorptiometry (DXA)
Fat mass | Baseline
  Fat mass using dual-energy x-ray absorptiometry (DXA)
Bone Mineral Density | Baseline
  Bone Mineral Density using dual-energy x-ray absorptiometry (DXA)
Appetite assessment | 4 hours after intervention
  Hunger, satiety, fullness, and prospective food consumption will be rated using a visual analog scales (VAS). A line of 20 cm is drawn from left to right on A4 paper starting at 0 cm with " not hungry at all" ending at 20 cm with "never been more hungry in my life". The subject mark somewhere in between according to his subjective feeling, The length is reported and indicates the degree of hunger, eg. the longer the line the more hunger. In general the longer to right the person marks the line, the stronger is the subjective felling within the given question
Ad libitum caloric intake | 4 hours after intervention
  Caloric intake will be determined by providing meal consisting of a hot pot of homogeneous pasta Bolognese (1,440 g, 1,912 kcal, 55 E percent carbohydrate, 30 E percent fat, 15 E percent protein; homogeneous composition) served with a glass of water of 150 ml 1 h after exercise. Participants will sit quietly on their own and are asked to eat until comfortably full/satiated and to drink all of the water. The duration of the meal is sat to 30 minutes
Gastric emptying | 4 hours after intervention
  Gastric emptying will be assessed by the participants drinking 100 ml in which 1,5 g paracetamol is dissolved. The Paracetamol concentration will be determined by Sandwich Electro-Chemiluminescence-Immunoassay (ECLIA)
Change in GLP1 | 4 hours after intervention
  Plasma GLP1 conc. using ELISA assay
Change in PYY | 4 hours after intervention
  Plasma PYY conc. using ELISA assay
Change in CCK | 4 hours after intervention
  Plasma CCK conc. using ELISA assay
Change in Glucose | 4 hours after intervention
  Plasma Glucose conc. using using sysmex XN
Change in Insulin | 4 hours after intervention
  Plasma insulin conc. using using sysmex XN
Change in C-peptide | 4 hours after intervention
  Plasma C-peptide conc. using using sysmex XN
Change in free fatty acids | 4 hours after intervention
  Plasma free fatty acids conc. using sysmex XN
Change in acetoacetate | 4 hours after intervention
  Plasma acetoacetate conc. using mass spectrometry
Change in betahydroxybutyrate | 4 hours after intervention
  Plasma betahydroxybutyrate conc. using mass spectrometry
Change in CRH | 4 hours after intervention
  Plasma CRH conc. using ELISA
Change in AVP | 4 hours after intervention
  Plasma AVP conc. using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Andreas K Ziegler, PhD, Principal Investigator — CFAS (Center For Physical Activity) Rigshospitalet; Jesper F Christensen, PhD, Principal Investigator — CFAS (Center For Physical Activity) Rigshospitalet; Claus Brandt, PhD, Principal Investigator — CFAS (Center For Physical Activity) Rigshospitalet
Locations (1):
- Center For Physical Activity (CFAS), Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amar, D., Lindholm, M. E., Norrbom, J., Wheeler, M. T., Rivas, M., & Ashley, E. A. (2020). Differential Response Trajectories to Acute Exercise in Blood and Muscle. SSRN Electronic Journal, 1-43. https://doi.org/10.2139/ssrn.3508810
- [Background] Bergstrom J. Percutaneous needle biopsy of skeletal muscle in physiological and clinical research. Scand J Clin Lab Invest. 1975 Nov;35(7):609-16. No abstract available. PMID 1108172
- [Background] Bigley AB, Rezvani K, Chew C, Sekine T, Pistillo M, Crucian B, Bollard CM, Simpson RJ. Acute exercise preferentially redeploys NK-cells with a highly-differentiated phenotype and augments cytotoxicity against lymphoma and multiple myeloma target cells. Brain Behav Immun. 2014 Jul;39:160-71. doi: 10.1016/j.bbi.2013.10.030. Epub 2013 Nov 5. PMID 24200514
- [Background] Chan CJ, Smyth MJ, Martinet L. Molecular mechanisms of natural killer cell activation in response to cellular stress. Cell Death Differ. 2014 Jan;21(1):5-14. doi: 10.1038/cdd.2013.26. Epub 2013 Apr 12. PMID 23579243
- [Background] Christensen JF, Simonsen C, Hojman P. Exercise Training in Cancer Control and Treatment. Compr Physiol. 2018 Dec 13;9(1):165-205. doi: 10.1002/cphy.c180016. PMID 30549018
- [Background] Dogra P, Rancan C, Ma W, Toth M, Senda T, Carpenter DJ, Kubota M, Matsumoto R, Thapa P, Szabo PA, Li Poon MM, Li J, Arakawa-Hoyt J, Shen Y, Fong L, Lanier LL, Farber DL. Tissue Determinants of Human NK Cell Development, Function, and Residence. Cell. 2020 Feb 20;180(4):749-763.e13. doi: 10.1016/j.cell.2020.01.022. Epub 2020 Feb 13. PMID 32059780
- [Background] Ghanemi A, St-Amand J. Interleukin-6 as a "metabolic hormone". Cytokine. 2018 Dec;112:132-136. doi: 10.1016/j.cyto.2018.06.034. Epub 2018 Jul 6. PMID 29983356
- [Background] Gjevestad GO, Holven KB, Ulven SM. Effects of Exercise on Gene Expression of Inflammatory Markers in Human Peripheral Blood Cells: A Systematic Review. Curr Cardiovasc Risk Rep. 2015;9(7):34. doi: 10.1007/s12170-015-0463-4. PMID 26005511
- [Background] Gupta P, Bigley AB, Markofski M, Laughlin M, LaVoy EC. Autologous serum collected 1 h post-exercise enhances natural killer cell cytotoxicity. Brain Behav Immun. 2018 Jul;71:81-92. doi: 10.1016/j.bbi.2018.04.007. Epub 2018 Apr 12. PMID 29656052
- [Background] Hanna J, Bechtel P, Zhai Y, Youssef F, McLachlan K, Mandelboim O. Novel insights on human NK cells' immunological modalities revealed by gene expression profiling. J Immunol. 2004 Dec 1;173(11):6547-63. doi: 10.4049/jimmunol.173.11.6547. PMID 15557145
- [Background] Kenfield SA, Stampfer MJ, Giovannucci E, Chan JM. Physical activity and survival after prostate cancer diagnosis in the health professionals follow-up study. J Clin Oncol. 2011 Feb 20;29(6):726-32. doi: 10.1200/JCO.2010.31.5226. Epub 2011 Jan 4. PMID 21205749
- [Background] Larrabee RC. Leucocytosis after violent Exercise. J Med Res. 1902 Jan;7(1):76-82. No abstract available. PMID 19971455
- [Background] Larsen SK, Gao Y, Basse PH. NK cells in the tumor microenvironment. Crit Rev Oncog. 2014;19(1-2):91-105. doi: 10.1615/critrevoncog.2014011142. PMID 24941376
- [Background] Lukaski HC. Soft tissue composition and bone mineral status: evaluation by dual-energy X-ray absorptiometry. J Nutr. 1993 Feb;123(2 Suppl):438-43. PMID 8429400
- [Background] Macpherson RE, Huber JS, Frendo-Cumbo S, Simpson JA, Wright DC. Adipose Tissue Insulin Action and IL-6 Signaling after Exercise in Obese Mice. Med Sci Sports Exerc. 2015 Oct;47(10):2034-42. doi: 10.1249/MSS.0000000000000660. PMID 25785928
- [Background] Meyerhardt JA, Giovannucci EL, Ogino S, Kirkner GJ, Chan AT, Willett W, Fuchs CS. Physical activity and male colorectal cancer survival. Arch Intern Med. 2009 Dec 14;169(22):2102-8. doi: 10.1001/archinternmed.2009.412. PMID 20008694
- [Background] Nieman DC, Miller AR, Henson DA, Warren BJ, Gusewitch G, Johnson RL, Davis JM, Butterworth DE, Nehlsen-Cannarella SL. Effects of high- vs moderate-intensity exercise on natural killer cell activity. Med Sci Sports Exerc. 1993 Oct;25(10):1126-34. PMID 8231757
- [Background] Ostrowski K, Rohde T, Asp S, Schjerling P, Pedersen BK. Pro- and anti-inflammatory cytokine balance in strenuous exercise in humans. J Physiol. 1999 Feb 15;515 ( Pt 1)(Pt 1):287-91. doi: 10.1111/j.1469-7793.1999.287ad.x. PMID 9925898
- [Background] Pedersen BK, Hoffman-Goetz L. Exercise and the immune system: regulation, integration, and adaptation. Physiol Rev. 2000 Jul;80(3):1055-81. doi: 10.1152/physrev.2000.80.3.1055. PMID 10893431
- [Background] Pedersen L, Idorn M, Olofsson GH, Lauenborg B, Nookaew I, Hansen RH, Johannesen HH, Becker JC, Pedersen KS, Dethlefsen C, Nielsen J, Gehl J, Pedersen BK, Thor Straten P, Hojman P. Voluntary Running Suppresses Tumor Growth through Epinephrine- and IL-6-Dependent NK Cell Mobilization and Redistribution. Cell Metab. 2016 Mar 8;23(3):554-62. doi: 10.1016/j.cmet.2016.01.011. Epub 2016 Feb 16. PMID 26895752
- [Background] Perez SA, Mahaira LG, Demirtzoglou FJ, Sotiropoulou PA, Ioannidis P, Iliopoulou EG, Gritzapis AD, Sotiriadou NN, Baxevanis CN, Papamichail M. A potential role for hydrocortisone in the positive regulation of IL-15-activated NK-cell proliferation and survival. Blood. 2005 Jul 1;106(1):158-66. doi: 10.1182/blood-2004-08-3232. Epub 2005 Mar 8. PMID 15755904
- [Background] Radom-Aizik S, Zaldivar F, Haddad F, Cooper DM. Impact of brief exercise on peripheral blood NK cell gene and microRNA expression in young adults. J Appl Physiol (1985). 2013 Mar 1;114(5):628-36. doi: 10.1152/japplphysiol.01341.2012. Epub 2013 Jan 3. PMID 23288554
- [Background] Rooney BV, Bigley AB, LaVoy EC, Laughlin M, Pedlar C, Simpson RJ. Lymphocytes and monocytes egress peripheral blood within minutes after cessation of steady state exercise: A detailed temporal analysis of leukocyte extravasation. Physiol Behav. 2018 Oct 1;194:260-267. doi: 10.1016/j.physbeh.2018.06.008. Epub 2018 Jun 7. PMID 29885920
- [Background] Schlahsa L, Jaimes Y, Blasczyk R, Figueiredo C. Granulocyte-colony-stimulatory factor: a strong inhibitor of natural killer cell function. Transfusion. 2011 Feb;51(2):293-305. doi: 10.1111/j.1537-2995.2010.02820.x. Epub 2010 Aug 16. PMID 20723170
- [Background] Smolen JS, Beaulieu A, Rubbert-Roth A, Ramos-Remus C, Rovensky J, Alecock E, Woodworth T, Alten R; OPTION Investigators. Effect of interleukin-6 receptor inhibition with tocilizumab in patients with rheumatoid arthritis (OPTION study): a double-blind, placebo-controlled, randomised trial. Lancet. 2008 Mar 22;371(9617):987-97. doi: 10.1016/S0140-6736(08)60453-5. PMID 18358926
- [Background] Wild CP, Weiderpass E, Stewart BW, editors. World Cancer Report: Cancer research for cancer prevention. Lyon (FR): International Agency for Research on Cancer; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK606505/ PMID 39432694
- [Background] Vivier E, Tomasello E, Baratin M, Walzer T, Ugolini S. Functions of natural killer cells. Nat Immunol. 2008 May;9(5):503-10. doi: 10.1038/ni1582. PMID 18425107
- [Background] Wang Y, Jacobs EJ, Gapstur SM, Maliniak ML, Gansler T, McCullough ML, Stevens VL, Patel AV. Recreational Physical Activity in Relation to Prostate Cancer-specific Mortality Among Men with Nonmetastatic Prostate Cancer. Eur Urol. 2017 Dec;72(6):931-939. doi: 10.1016/j.eururo.2017.06.037. Epub 2017 Jul 12. PMID 28711382
- [Background] Weber MM, Michl P, Auernhammer CJ, Engelhardt D. Interleukin-3 and interleukin-6 stimulate cortisol secretion from adult human adrenocortical cells. Endocrinology. 1997 May;138(5):2207-10. doi: 10.1210/endo.138.5.5239. PMID 9112422
- [Background] Wendt K, Wilk E, Buyny S, Buer J, Schmidt RE, Jacobs R. Gene and protein characteristics reflect functional diversity of CD56dim and CD56bright NK cells. J Leukoc Biol. 2006 Dec;80(6):1529-41. doi: 10.1189/jlb.0306191. Epub 2006 Sep 11. PMID 16966385
- [Background] Wu J, Lanier LL. Natural killer cells and cancer. Adv Cancer Res. 2003;90:127-56. doi: 10.1016/s0065-230x(03)90004-2. PMID 14710949
- [Background] Yamada M, Suzuki K, Kudo S, Totsuka M, Nakaji S, Sugawara K. Raised plasma G-CSF and IL-6 after exercise may play a role in neutrophil mobilization into the circulation. J Appl Physiol (1985). 2002 May;92(5):1789-94. doi: 10.1152/japplphysiol.00629.2001. PMID 11960925
- [Background] Zimmer P, Schenk A, Kieven M, Holthaus M, Lehmann J, Lovenich L, Bloch W. Exercise induced alterations in NK-cell cytotoxicity - methodological issues and future perspectives. Exerc Immunol Rev. 2017;23:66-81. PMID 28230531
- [Background] Dorling J, Broom DR, Burns SF, Clayton DJ, Deighton K, James LJ, King JA, Miyashita M, Thackray AE, Batterham RL, Stensel DJ. Acute and Chronic Effects of Exercise on Appetite, Energy Intake, and Appetite-Related Hormones: The Modulating Effect of Adiposity, Sex, and Habitual Physical Activity. Nutrients. 2018 Aug 22;10(9):1140. doi: 10.3390/nu10091140. PMID 30131457
- [Background] Steensberg A, van Hall G, Osada T, Sacchetti M, Saltin B, Klarlund Pedersen B. Production of interleukin-6 in contracting human skeletal muscles can account for the exercise-induced increase in plasma interleukin-6. J Physiol. 2000 Nov 15;529 Pt 1(Pt 1):237-42. doi: 10.1111/j.1469-7793.2000.00237.x. PMID 11080265
- [Background] Dantzer R. Cytokine-induced sickness behavior: mechanisms and implications. Ann N Y Acad Sci. 2001 Mar;933:222-34. doi: 10.1111/j.1749-6632.2001.tb05827.x. PMID 12000023
- [Background] van Gameren MM, Willemse PH, Mulder NH, Limburg PC, Groen HJ, Vellenga E, de Vries EG. Effects of recombinant human interleukin-6 in cancer patients: a phase I-II study. Blood. 1994 Sep 1;84(5):1434-41. PMID 8068939
- [Background] Timper K, Denson JL, Steculorum SM, Heilinger C, Engstrom-Ruud L, Wunderlich CM, Rose-John S, Wunderlich FT, Bruning JC. IL-6 Improves Energy and Glucose Homeostasis in Obesity via Enhanced Central IL-6 trans-Signaling. Cell Rep. 2017 Apr 11;19(2):267-280. doi: 10.1016/j.celrep.2017.03.043. PMID 28402851
- [Background] Lang Lehrskov L, Lyngbaek MP, Soederlund L, Legaard GE, Ehses JA, Heywood SE, Wewer Albrechtsen NJ, Holst JJ, Karstoft K, Pedersen BK, Ellingsgaard H. Interleukin-6 Delays Gastric Emptying in Humans with Direct Effects on Glycemic Control. Cell Metab. 2018 Jun 5;27(6):1201-1211.e3. doi: 10.1016/j.cmet.2018.04.008. Epub 2018 May 3. PMID 29731416
- [Background] Ellingsgaard H, Seelig E, Timper K, Coslovsky M, Soederlund L, Lyngbaek MP, Wewer Albrechtsen NJ, Schmidt-Trucksass A, Hanssen H, Frey WO, Karstoft K, Pedersen BK, Boni-Schnetzler M, Donath MY. GLP-1 secretion is regulated by IL-6 signalling: a randomised, placebo-controlled study. Diabetologia. 2020 Feb;63(2):362-373. doi: 10.1007/s00125-019-05045-y. Epub 2019 Dec 3. PMID 31796986
- [Background] Begg DP, Woods SC. The endocrinology of food intake. Nat Rev Endocrinol. 2013 Oct;9(10):584-97. doi: 10.1038/nrendo.2013.136. Epub 2013 Jul 23. PMID 23877425
- [Background] Medhus AW, Sandstad O, Bredesen J, Husebye E. Delay of gastric emptying by duodenal intubation: sensitive measurement of gastric emptying by the paracetamol absorption test. Aliment Pharmacol Ther. 1999 May;13(5):609-20. doi: 10.1046/j.1365-2036.1999.00519.x. PMID 10233184